CLINICAL TRIAL: NCT05495997
Title: Effects of Cognitive Training on Everyday Cognitive and Brain Function in Parkinson's Disease
Brief Title: Cognitive Training in Parkinson's Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2000033352; R56NS129540 (NIH)
Record Dates: First submitted 2022-08-08; First posted 2022-08-10 (Actual); Results first posted 2025-07-17 (Actual); Last update posted 2025-08-11 (Actual); Status verified 2025-07

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mental Imagery (Experimental)
  Interventions: Behavioral: Mental Imagery Training
- Psychoeducation (Active Comparator)
  Interventions: Behavioral: Psychoeducation

INTERVENTIONS:
Behavioral: Mental Imagery Training — Participants will practice mental imagery of everyday tasks daily for 6 weeks.
  Arms: Mental Imagery
Behavioral: Psychoeducation — Participants will receive psychoeducation on cognition and brain health.
  Arms: Psychoeducation

SUMMARY:
The purpose of this research study is to determine whether cognitive training will improve cognitive and brain functions in people with Parkinson's Disease (PD) during activities of daily living using cognitive evaluations and magnetic resonance imaging (MRI).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of idiopathic PD
* Age ≥ 40 years
* Expected to be on a stable dopaminergic medication regimen throughout the study period

Exclusion Criteria:

* Non-English speaking
* Pregnancy
* Breastfeeding
* Excessive alcohol consumption (> 7 drinks per week for women, > 14 drinks per week for men) or illicit substance use
* History of a neurological disorder such as a brain tumor, stroke, central nervous system infection, multiple sclerosis, movement disorder (other than PD), or seizures
* History of schizophrenia, bipolar disorder, attention deficit disorder, or obsessive-compulsive disorder
* History of head injury with loss of consciousness longer than a few minutes
* Metallic surgical implants or traumatically implanted metallic foreign bodies
* Inability to lie flat for about an hour in the MRI scanner
* Discomfort being in small, enclosed spaces
* Dementia at screening (Montreal Cognitive Assessment score < 21/30)
* Cognitive problems in activities of daily living suggestive of more than mild cognitive impairment (PD Cognitive Functional Rating Scale > 4)
* Mild cognitive impairment according to the Movement Disorders Society (MDS) Level II comprehensive assessment criteria (> 1.5 standard deviations below the norm in two tests in a single cognitive domain or in one test in two separate cognitive domains, with the exception that the executive domain scores can be up to 2 standard deviations below the norm)
* Hoehn & Yahr stage > 3 (i.e., able to stand and walk, but not fully independent)
* Focal neurological findings on exam that suggest cerebral pathology other than that associated with parkinsonism
* Motor symptoms that could potentially introduce too much motion artifact in the imaging data (e.g., MDS-Unified PD Rating Scale resting tremor score > 2 in limbs, head/chin tremor, or more than mild dyskinesia by history or exam)

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2023-01-13 (Actual); Primary Completion 2024-09-18 (Actual); Study Completion 2024-09-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sule Tinaz, MD, PhD, Principal Investigator — Yale University
Locations (1):
- Yale School of Medicine, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: Yes
This study will produce unique clinical, cognitive, behavioral, and imaging datasets obtained from subjects with mild-to-moderate Parkinson's disease at baseline and at two time points - immediate and delayed - post-intervention. The de-identified datasets will be made available for research purposes to qualified individuals within the scientific community upon request.
Supporting Information: Study Protocol, SAP, CSR, Analytic Code
Time Frame: Beginning 9 months and ending 36 months following article publication.

REFERENCES:
- [Derived] Cherry J, Nelson AM, Robinson LA, Goldstein J, Vives-Rodriguez A, Sharp E, Tinaz S. Feasibility and potential effects of mental imagery training on subjective cognitive function and brain connectivity in people with Parkinson's disease: A randomized pilot trial. Neuropsychol Rehabil. 2026 Jan 3:1-28. doi: 10.1080/09602011.2025.2608220. Online ahead of print. PMID 41482867
- [Derived] Cherry J, Nelson AM, Robinson LA, Goldstein J, Vives-Rodriguez A, Sharp E, Tinaz S. Effects of mental imagery training on cognitive function and brain connectivity in people with Parkinson's disease: A randomized pilot trial. medRxiv [Preprint]. 2025 Mar 15:2025.03.14.25324001. doi: 10.1101/2025.03.14.25324001. PMID 40162247

RESULTS

PARTICIPANT FLOW:
Groups:
- Mental Imagery: Participants will practice mental imagery of everyday tasks daily for 6 weeks.
Period: Overall Study
Arm/Group | Mental Imagery | Psychoeducation
Started | 15 | 15
Completed 18 Week Follow up Cognitive Tests | 15 | 13
Completed 18 Week Follow up fMRI | 15 | 12
Completed | 15 | 13
Not Completed | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Mental Imagery | Psychoeducation | Total
Number analyzed (Participants) | 15 | 15 | 30
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.6 (8.6) | 67.5 (7.7) | 67.6 (8.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 3 | 7
  Male | 11 | 12 | 23
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 0 | 2
  Not Hispanic or Latino | 13 | 15 | 28
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 12 | 14 | 26
  More than one race | 2 | 0 | 2
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: Participants]
  United States | 15 | 15 | 30
Years of Education [Mean (Standard Deviation); unit: years] | 17.1 (1.9) | 18.3 (1.8) | 17.7 (1.9)

OUTCOME MEASURES:

1. Primary Outcome: Change in Quality of Life in Neurological Disorders Cognitive Function Version 2 (Neuro-QoL CF v2) T-scores at 6 Weeks
Description: Neuro-QoL CF v2 measures self-reported levels of cognitive functioning. Raw scores are converted to standardized T-scores (mean of 50 with a standard deviation of 10). Increase in T-scores from baseline indicates improvement in everyday cognitive functioning.
Time Frame: Baseline and 6 weeks
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | Mental Imagery | Psychoeducation
Number analyzed (Participants) | 15 | 15
T-score
  Baseline | 49.9 (7.2) | 49.1 (8.4)
  6 weeks | 50 (7.2) | 45.9 (5.1)
Statistical Analysis 1: Comparison: Mental Imagery vs Psychoeducation; Mental Imagery Group (PD-MI) compared to Psychoeducation Control Group (PD-Con) at 6 weeks compared to baseline (group-by-time interaction); Test type: Superiority; p = 0.015, ANCOVA

2. Primary Outcome: Change in Neuro-QoL CF v2 T-scores at 18 Weeks
Description: as for outcome 1
Time Frame: 18 weeks
Population: 15 in the Mental Imagery and 13 in the Psychoeducation group completed 18-week assessments.
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | Mental Imagery | Psychoeducation
Number analyzed (Participants) | 15 | 13
T-score
  Baseline | 49.9 (7.2) | 49.1 (8.4)
  18 weeks | 49.4 (7.4) | 46.9 (6.1)
Statistical Analysis 1: Comparison: Mental Imagery vs Psychoeducation; Mental Imagery Group (PD-MI) compared to Psychoeducation Control Group (PD-Con) at 18 weeks compared to baseline (group-by-time interaction); Test type: Superiority; p = 0.993, ANCOVA

3. Secondary Outcome: Change in Composite Executive Function T-scores at 6 Weeks
Description: T-scores (mean of 50 with a standard deviation of 10) of executive function tests (i.e., Stroop, F-A-S letter fluency, and Trail Making B tests) were averaged to obtain a composite executive function score for each subject. Higher scores indicate better executive function.
Time Frame: 6 weeks
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | Mental Imagery | Psychoeducation
Number analyzed (Participants) | 15 | 15
T-score
  Baseline | 53.1 (7.9) | 48.7 (7.4)
  6 weeks | 54.7 (8.2) | 51 (9.5)
Statistical Analysis 1: Comparison: Mental Imagery vs Psychoeducation; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.517, ANCOVA

4. Secondary Outcome: Change in Composite Executive Function T-scores at 18 Weeks
Description: as for outcome 3
Time Frame: 18 weeks
Population: 15 in the Mental Imagery group and 13 in the Psychoeducation group completed 18-week assessments
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | Mental Imagery | Psychoeducation
Number analyzed (Participants) | 15 | 13
T-score
  Baseline | 53.1 (7.9) | 48.7 (7.4)
  18 weeks | 55.1 (9.6) | 49.5 (7.8)
Statistical Analysis 1: Comparison: Mental Imagery vs Psychoeducation; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.817, ANCOVA

ADVERSE EVENTS:
Time Frame: 18 weeks
Arm/Group | Mental Imagery | Psychoeducation
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/15
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/15
Other Adverse Events (participants affected / at risk) | 0/15 | 0/15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-09-28): https://cdn.clinicaltrials.gov/large-docs/97/NCT05495997/Prot_SAP_000.pdf
  • Informed Consent Form (2022-11-23): https://cdn.clinicaltrials.gov/large-docs/97/NCT05495997/ICF_001.pdf